CLINICAL TRIAL: NCT00322946
Title: Phase 1 Study of the Safety and Immunogenicity of rDEN4delta30-4995, a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 4
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN4delta30-4995) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 221; WIRB Protocol Number 20061807
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2008-11

CONDITIONS: Dengue
Keywords: Dengue Fever; Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): One subcutaneous vaccination with rDEN4delta30-4995 vaccine (10^5 PFU dose) into the deltoid region of either arm.
  Interventions: Biological: rDEN4delta30-4995
- 2 (Experimental): One subcutaneous vaccination with rDEN4delta30-4995 vaccine (10^3 PFU dose) into the deltoid region of either arm. This arm will enroll after Arm 1.
  Interventions: Biological: rDEN4delta30-4995
- 3 (Experimental): One subcutaneous vaccination with rDEN4delta30-4995 vaccine (10^1 PFU dose) into the deltoid region of either arm. This arm will enroll after Arms 1 and 2.
  Interventions: Biological: rDEN4delta30-4995
- 4 (Placebo Comparator): One subcutaneous vaccination with placebo into the deltoid region of either arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN4delta30-4995 — Live attenuated rDEN4delta30-4995 vaccine (one of three doses)
  Arms: 1; 2; 3
Biological: Placebo — Placebo for rDEN4delta30-4995
  Arms: 4

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to evaluate the safety and immune response to the dengue vaccine DEN4delta30-4995 in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses account for more than 50 million cases of dengue fever and a half million cases of the more severe disease, dengue hemorrhagic fever/dengue shock syndrome. Infection with dengue viruses is the leading cause of hospitalization and death in children in at least eight Asian countries. The goal of producing a vaccine against dengue fever is to induce a long-lived antibody response against all four dengue serotypes. The rDEN4delta30-4995 vaccine candidate is a live attenuated recombinant virus derived from rDEN4delta30 for protection against dengue virus serotype 4. The purpose of this study is to evaluate the safety, reactogenicity, and immunogenicity of rDEN4delta30-4995 in healthy adults.

This study will last 180 days (6 months). Participants in Cohort 1 will be randomly assigned to receive the highest dose of rDEN4delta30 or placebo at study entry. Participants in Cohort 2 will be randomly assigned to receive a lower dose of rDEN4delta30 or placebo. Participants in Cohort 3 will be randomly assigned to receive the lowest dose of rDEN4delta30 or placebo. Cohorts 2 and 3 will begin after a safety review of all participants in the previous cohort.

After initial vaccination, participants in Cohort 1 will be followed every other day for the first 16 days of the study, monitoring their temperature three times a day through Day 16 and recording these measurements in a diary. After Day 16, study visits will occur on Days 21, 28, 42, and 180 and will include a physical exam and blood collection. Some participants will also be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and non-pregnant females between 18 and 50 years of age
* Good general health
* Available for the duration of the study
* Willing to use acceptable methods of contraception for the duration of the study

Exclusion Criteria:

* Significant neurologic, cardiac, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, may interfere with the study
* Significant laboratory abnormalities
* Medical, work, or family problems as a result of alcohol or illegal drug use within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Severe asthma
* HIV-1 serotype infected
* Hepatitis C virus (HCV) infected
* Hepatitis B surface antigen positive
* Immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive medications within 2 weeks prior to study entry. Individuals using topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Absence of spleen
* Blood products within 6 months prior to study entry
* Previous dengue virus or other flavivirus (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus) infection
* Prior receipt of yellow fever or dengue vaccine (licensed or experimental)
* Plans to travel to an area where dengue infection is common
* Received an investigational agent within 30 days prior to study entry
* Other condition that, in the opinion of the investigator, would affect participation in the study
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse events, graded by severity for each dose | Throughout study
Immunogenicity of the rDEN4delta30-4995 vaccine against DEN4 virus by measurement of plaque reduction neutralization titers (PRNT) | At Days 28 and 42

SECONDARY OUTCOMES:
Durability of antibody responses to DEN4 virus | At Month 6
Frequency, quantity, and duration of viremia in each dose cohort studied based on the mean peak viremia, mean day onset of viremia, and mean duration of viremia of each dose cohort | Throughout study
Number of vaccinees infected with the rDEN4delta30-4995 chimeric vaccine | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health
Locations (1):
- Vanderbilt University School of Medicine, Nashville, Tennessee, United States

REFERENCES:
- [Background] Bhamarapravati N, Sutee Y. Live attenuated tetravalent dengue vaccine. Vaccine. 2000 May 26;18 Suppl 2:44-7. doi: 10.1016/s0264-410x(00)00040-2. PMID 10821973
- [Background] Blaney JE Jr, Durbin AP, Murphy BR, Whitehead SS. Development of a live attenuated dengue virus vaccine using reverse genetics. Viral Immunol. 2006 Spring;19(1):10-32. doi: 10.1089/vim.2006.19.10. PMID 16553547
- [Background] Durbin AP, Whitehead SS, McArthur J, Perreault JR, Blaney JE Jr, Thumar B, Murphy BR, Karron RA. rDEN4delta30, a live attenuated dengue virus type 4 vaccine candidate, is safe, immunogenic, and highly infectious in healthy adult volunteers. J Infect Dis. 2005 Mar 1;191(5):710-8. doi: 10.1086/427780. Epub 2005 Jan 27. PMID 15688284
- [Background] Durbin AP, Karron RA, Sun W, Vaughn DW, Reynolds MJ, Perreault JR, Thumar B, Men R, Lai CJ, Elkins WR, Chanock RM, Murphy BR, Whitehead SS. Attenuation and immunogenicity in humans of a live dengue virus type-4 vaccine candidate with a 30 nucleotide deletion in its 3'-untranslated region. Am J Trop Med Hyg. 2001 Nov;65(5):405-13. doi: 10.4269/ajtmh.2001.65.405. PMID 11716091